CLINICAL TRIAL: NCT01002053
Title: Can Ultrasound Predict Nerve Injury Following Posterior Tibial Nerve Block in Patients With Peripheral Neuropathy?
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: UHN 09-0803-AE
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2011-11

CONDITIONS: Diabetic Neuropathy
Keywords: diabetes; neuropathy; ankle block; regional anesthesia; ultrasound; nerve localization; Nerve localization in patients undergoing foot surgery and having ankle block
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diabetics with peripheral neuropathy: Patients with diabetes and peripheral neuropathy.
  Interventions: Procedure: Nerve conduction study and Ultrasound of the PTN

INTERVENTIONS:
Procedure: Nerve conduction study and Ultrasound of the PTN — Nerve Conduction studies and ultrasound of PTN will be performed to the patient before the operation and 8 weeks postoperatively.

SUMMARY:
The use of regional anesthesia for nerve block in diabetic patients with peripheral neuropathy is currently made on a case-by-case basis, also remains underlying uncertainty regarding the preferred technique and the likelihood of block-related nerve injury. For this many diabetic patients with otherwise healthy nerves may receive general anesthesia instead of regional anesthesia, thus giving up the benefits associated with the latter technique, including a decrease in health complications and superior analgesia following the operation. Ultrasound is used to identify the target nerve and guide needle insertion for nerve blocks, may be a useful tool to detect the presence and severity of neuropathy prior to block placement, a recent study demonstrated a statistically significant increase in the sonographic cross-sectional area of the posterior tibial nerve (PTN) in all diabetic patients who had abnormal motor transmission on nerve conduction studies. For regional anesthesiologists, the ultimate goal of detecting peripheral neuropathy and in particular, diabetic neuropathy by US is to avoid nerve injury. To do so, the association between US-detected diabetic neuropathy and block-related nerve damage must be first established, hence the purpose of this study. We aim to examine whether the cross-sectional area of PTN as assessed by preoperative US can predict nerve injury as assessed by worsening nerve conduction studies following PTN block inpatients scheduled to receive an ankle block. A further subgroup analysis will be performed in diabetic patients.

We hypothesize that the cross sectional area of the PTN will correlate with motor conduction velocity on nerve conduction studies (NCS) following PTN block in patients with peripheral neuropathy. All eligible patients will undergo NCS to confirm or exclude distal neuropathy. Patients without neuropathy will be excluded from further participation in this study. Also excluded will be diabetic patients with neuropathy caused by genetic, metabolic and inflammatory diseases as well as toxic agents and drug induced. A systematic US examination of the PTN will be performed for all patients. After Block administration at surgery day the block successes will be assessed and for the purposes of the present study, patients in whom the block was not successful will be excluded from further intervention and data analyses. Eight weeks after surgery, all study patients will return to hospital for repeat NCS and US.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing PTN block for foot surgery
* Type I diabetic patients (diagnosed more than 5 years), and II diabetic patients with demonstrated peripheral neuropathy
* ASA I-III

Exclusion Criteria:

* Non-diabetic neuropathy caused by genetic, metabolic and inflammatory diseases as well as toxic agents and drug induced (e.g. chemotherapy agents)
* Psychiatric history
* Allergy to local anesthetics

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic and non-diabetic patients undergoing foot surgery involving regional anesthesia/nerve blockade.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-02; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Interval worsening of the severity of neuropathy | 8 weeks

SECONDARY OUTCOMES:
New functional neuropathy defined as any new sensory or motor deficit compared to preoperatively. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Riazi, MD, MSc, FRCPC, Principal Investigator — University Health Network - University of Toronto
Locations (1):
- Toronto Western Hospital, University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Background] Upton AR, McComas AJ. The double crush in nerve entrapment syndromes. Lancet. 1973 Aug 18;2(7825):359-62. doi: 10.1016/s0140-6736(73)93196-6. No abstract available. PMID 4124532
- [Background] Blumenthal S, Borgeat A, Maurer K, Beck-Schimmer B, Kliesch U, Marquardt M, Urech J. Preexisting subclinical neuropathy as a risk factor for nerve injury after continuous ropivacaine administration through a femoral nerve catheter. Anesthesiology. 2006 Nov;105(5):1053-6. doi: 10.1097/00000542-200611000-00028. No abstract available. PMID 17065901
- [Background] Zochodne DW. Diabetic polyneuropathy: an update. Curr Opin Neurol. 2008 Oct;21(5):527-33. doi: 10.1097/WCO.0b013e32830b84cb. PMID 18769245
- [Background] Dyck PJ, Karnes JL, O'Brien PC, Litchy WJ, Low PA, Melton LJ 3rd. The Rochester Diabetic Neuropathy Study: reassessment of tests and criteria for diagnosis and staged severity. Neurology. 1992 Jun;42(6):1164-70. doi: 10.1212/wnl.42.6.1164. PMID 1603343
- [Background] Kalichman MW, Calcutt NA. Local anesthetic-induced conduction block and nerve fiber injury in streptozotocin-diabetic rats. Anesthesiology. 1992 Nov;77(5):941-7. doi: 10.1097/00000542-199211000-00017. PMID 1443749
- [Background] Hebl JR, Kopp SL, Schroeder DR, Horlocker TT. Neurologic complications after neuraxial anesthesia or analgesia in patients with preexisting peripheral sensorimotor neuropathy or diabetic polyneuropathy. Anesth Analg. 2006 Nov;103(5):1294-9. doi: 10.1213/01.ane.0000243384.75713.df. PMID 17056972
- [Background] Kroin JS, Buvanendran A, Williams DK, Wagenaar B, Moric M, Tuman KJ, Kerns JM. Local anesthetic sciatic nerve block and nerve fiber damage in diabetic rats. Reg Anesth Pain Med. 2010 Jul-Aug;35(4):343-50. doi: 10.1097/aap.0b013e3181e82df0. PMID 20607875
- [Background] Ballantyne JC, Carr DB, deFerranti S, Suarez T, Lau J, Chalmers TC, Angelillo IF, Mosteller F. The comparative effects of postoperative analgesic therapies on pulmonary outcome: cumulative meta-analyses of randomized, controlled trials. Anesth Analg. 1998 Mar;86(3):598-612. doi: 10.1097/00000539-199803000-00032. PMID 9495424
- [Background] Urwin SC, Parker MJ, Griffiths R. General versus regional anaesthesia for hip fracture surgery: a meta-analysis of randomized trials. Br J Anaesth. 2000 Apr;84(4):450-5. doi: 10.1093/oxfordjournals.bja.a013468. PMID 10823094
- [Background] Hadzic A, Arliss J, Kerimoglu B, Karaca PE, Yufa M, Claudio RE, Vloka JD, Rosenquist R, Santos AC, Thys DM. A comparison of infraclavicular nerve block versus general anesthesia for hand and wrist day-case surgeries. Anesthesiology. 2004 Jul;101(1):127-32. doi: 10.1097/00000542-200407000-00020. PMID 15220781
- [Background] Chan VW, Peng PW, Kaszas Z, Middleton WJ, Muni R, Anastakis DG, Graham BA. A comparative study of general anesthesia, intravenous regional anesthesia, and axillary block for outpatient hand surgery: clinical outcome and cost analysis. Anesth Analg. 2001 Nov;93(5):1181-4. doi: 10.1097/00000539-200111000-00025. PMID 11682392
- [Background] Alshami AM, Cairns CW, Wylie BK, Souvlis T, Coppieters MW. Reliability and size of the measurement error when determining the cross-sectional area of the tibial nerve at the tarsal tunnel with ultrasonography. Ultrasound Med Biol. 2009 Jul;35(7):1098-102. doi: 10.1016/j.ultrasmedbio.2009.01.011. Epub 2009 May 7. PMID 19427097
- [Background] Cartwright MS, Passmore LV, Yoon JS, Brown ME, Caress JB, Walker FO. Cross-sectional area reference values for nerve ultrasonography. Muscle Nerve. 2008 May;37(5):566-71. doi: 10.1002/mus.21009. PMID 18351581
- [Background] Lee D, Dauphinee DM. Morphological and functional changes in the diabetic peripheral nerve: using diagnostic ultrasound and neurosensory testing to select candidates for nerve decompression. J Am Podiatr Med Assoc. 2005 Sep-Oct;95(5):433-7. doi: 10.7547/0950433. PMID 16166459
- [Background] Vijayan J, Therimadasamy AK, Teoh HL, Chan YC, Wilder-Smith EP. Sonography as an aid to neurophysiological studies in diagnosing tarsal tunnel syndrome. Am J Phys Med Rehabil. 2009 Jun;88(6):500-1. doi: 10.1097/PHM.0b013e3181a5b94b. PMID 19454856
- [Background] Watanabe T, Ito H, Morita A, Uno Y, Nishimura T, Kawase H, Kato Y, Matsuoka T, Takeda J, Seishima M. Sonographic evaluation of the median nerve in diabetic patients: comparison with nerve conduction studies. J Ultrasound Med. 2009 Jun;28(6):727-34. doi: 10.7863/jum.2009.28.6.727. PMID 19470812
- [Background] Watanabe T, Ito H, Sekine A, Katano Y, Nishimura T, Kato Y, Takeda J, Seishima M, Matsuoka T. Sonographic evaluation of the peripheral nerve in diabetic patients: the relationship between nerve conduction studies, echo intensity, and cross-sectional area. J Ultrasound Med. 2010 May;29(5):697-708. doi: 10.7863/jum.2010.29.5.697. PMID 20427781
- [Background] Harati Y. Diabetic neuropathies: unanswered questions. Neurol Clin. 2007 Feb;25(1):303-17. doi: 10.1016/j.ncl.2007.01.002. PMID 17324729
- [Background] Misur I, Zarkovic K, Barada A, Batelja L, Milicevic Z, Turk Z. Advanced glycation endproducts in peripheral nerve in type 2 diabetes with neuropathy. Acta Diabetol. 2004 Dec;41(4):158-66. doi: 10.1007/s00592-004-0160-0. PMID 15660198
- [Background] Partanen J, Niskanen L, Lehtinen J, Mervaala E, Siitonen O, Uusitupa M. Natural history of peripheral neuropathy in patients with non-insulin-dependent diabetes mellitus. N Engl J Med. 1995 Jul 13;333(2):89-94. doi: 10.1056/NEJM199507133330203. PMID 7777034
- [Background] Perkins BA, Bril V. Diabetic neuropathy: a review emphasizing diagnostic methods. Clin Neurophysiol. 2003 Jul;114(7):1167-75. doi: 10.1016/s1388-2457(03)00025-7. PMID 12842711
- [Background] Vinik AI, Bril V, Litchy WJ, Price KL, Bastyr EJ 3rd; MBBQ Study Group. Sural sensory action potential identifies diabetic peripheral neuropathy responders to therapy. Muscle Nerve. 2005 Nov;32(5):619-25. doi: 10.1002/mus.20423. PMID 16116628
- [Background] Olaleye D, Perkins BA, Bril V. Evaluation of three screening tests and a risk assessment model for diagnosing peripheral neuropathy in the diabetes clinic. Diabetes Res Clin Pract. 2001 Nov;54(2):115-28. doi: 10.1016/s0168-8227(01)00278-9. PMID 11640995
- [Background] Yesildag A, Kutluhan S, Sengul N, Koyuncuoglu HR, Oyar O, Guler K, Gulsoy UK. The role of ultrasonographic measurements of the median nerve in the diagnosis of carpal tunnel syndrome. Clin Radiol. 2004 Oct;59(10):910-5. doi: 10.1016/j.crad.2004.03.020. PMID 15451351